CLINICAL TRIAL: NCT04035083
Title: Evaluation of Post-operative Pain and Bacterial Reduction Following Laser Activated Irrigation Versus Passive Ultrasonic Irrigation in Necrotic Single Rooted Teeth: A Randomized Clinical Trial
Brief Title: Laser Activated Irrigation Versus Passive Ultrasonic Irrigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ayman Abo El Enin Ahmed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAI_PUI
Record Dates: First submitted 2019-07-19; First posted 2019-07-29 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Pulp Necroses
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser activated irrigation (Experimental): Laser activated irrigation of sodium hypochlorite using a 980 nm diode laser device
  Interventions: Device: Laser activated irrigation
- Passive ultrasonic irrigation (Active Comparator): passive ultrasonic irrigation of sodium hypochlorite using an ultrasonic laser device
  Interventions: Device: Passive ultrasonic irrigation

INTERVENTIONS:
Device: Laser activated irrigation — Diode laser at 980 nm, power of 1.5W, for 5 seconds inside the canal along with sodium hypochlorite, repeated 4 times with a gap of 10 seconds in between
  Arms: Laser activated irrigation
Device: Passive ultrasonic irrigation — ultrasonic activation inside the canal for 1 min
  Arms: Passive ultrasonic irrigation

SUMMARY:
assessment of bacterial reduction and post-operative pain following Laser activated irrigation using sodium hypochlorite and a 980 nm diode laser device as an adjunct to conventional root canal treatment, and comparing it with passive ultrasonic irrigation using sodium hypochlorite and an ultrasonic device in patients with single rooted asymptomatic necrotic teeth.

DETAILED DESCRIPTION:
After thorough diagnosis and recording of the patient's perceived preoperative pain using the numeric rating scale (NRS), which should be zero. Patients with single rooted necrotic teeth will be randomly divided into two groups for endodontic treatment in a single visit:

Group LAI (in which laser activated irrigation will be done) and group PUI (in which passive ultrasonic irrigation will be done).

The teeth are anesthetized and isolation is done. the clamp, tooth crown and rubber dam are disinfected using 2.5% sodium hypochlorite and 30% hydrogen peroxide then sodium thiosulphate to neutralize their effects.

Removal of caries and defective restorations is done, followed by access cavity preparation using round burs and fine tapered stones. then the first microbiological sample is taken using paper points. Afterwards root canal preparation is done using Protaper Next files and irrigation is done using 2.5% sodium hypochlorite and a 30 -gauge side vented needle.

After chemomechanical preparation of the canal, the second microbiological sample is taken, afterwards the canals are filled with sodium hypochlorite and according to the group, the following is done:

In group LAI: the 200 micrometer fibre of the diode laser device enters the root canal and the device is activated at a setting of 980 nm and 1.5 Watts for 5 seconds, repeated 4 times with a 10 seconds gap in between.

In group PUI: the ultrasonic device is activated inside the canal using a passive non cutting tip and kept activated for 1 minute.

Then, irrigation with saline solution is done then the third microbiological sample is taken, afterwards obturation is done and temporization. the patient is referred to the restorative dentistry clinic to complete the restoration of his tooth.

The patient is instructed to record his pain at 6,12,24 and 48 hours postoperatively and the microbiological samples are analyzed

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Patients with necrotic pulp in single rooted teeth with:

  * Closed apex.
  * Associated with or without periapical radiolucency.
  * No response of vital pulp with the electric pulp tester.
* Healthy dental and periodontal status.
* Positive patients' acceptance for participation in the study.

Exclusion Criteria i. Patients on medication for chronic pain. ii. Patients with pre-operative pain. iii. Patients having significant systemic disorders. iv. Patients with two or more adjacent teeth requiring root canal therapy. v. Patients who had received antibiotics in the last month. vi. Teeth that have:

* Vital pulp tissues.
* Association with swelling or fistulous tract.
* Acute peri-apical abscess.
* Greater than grade I mobility.
* Pocket depth greater than 5mm.
* No possible restorability.
* Previous endodontic treatment.
* Open apex.
* Extra coronal restorations.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain 6 hours post-operatively: NRS | 6 hours after endodontic treatment
  Pain perceived by the patient using the 11-point numeric rating scale (NRS) with ranges from zero to 10 (zero meaning no pain, 1-3 means mild pain, 4-7 means moderate pain, 8-10 means severe pain with 10 being the highest pain imaginable)
Post-operative pain 12 hours post-operatively: NRS | 12 hours after endodontic treatment
  Pain perceived by the patient using the 11-point numeric rating scale (NRS) with ranges from zero to 10 (zero meaning no pain, 1-3 means mild pain, 4-7 means moderate pain, 8-10 means severe pain with 10 being the highest pain imaginable)
Post-operative pain 24 hours post-operatively: NRS | 24 hours after endodontic treatment
  Pain perceived by the patient using the 11-point numeric rating scale (NRS) with ranges from zero to 10 (zero meaning no pain, 1-3 means mild pain, 4-7 means moderate pain, 8-10 means severe pain with 10 being the highest pain imaginable)
Post-operative pain 48 hours post-operatively: NRS | 48 hours after endodontic treatment
  Pain perceived by the patient using the 11-point numeric rating scale (NRS) with ranges from zero to 10 (zero meaning no pain, 1-3 means mild pain, 4-7 means moderate pain, 8-10 means severe pain with 10 being the highest pain imaginable)

SECONDARY OUTCOMES:
change in intracanal bacterial flora count | 48 hours after endodontic treatment
  bacterial cultures made from microbiological samples taken at different stages of the endodontic treatment. The bacteria will be counted as colony forming units (CFUs). There are three samples that are taken during the endodontic treatment : S1: After Access cavity preparation. S2: After chemomechanical preparation S3: After using the intervention or control. The CFUs will be counted in the culture obtained from each sample then a comparison will be made between the intervention and control groups regarding the difference in the number of CFUs in S2 between S3

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Gawdat, PhD, Study Director — central evidence based dentistry committee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dagher J, El Feghali R, Parker S, Benedicenti S, Zogheib C. Postoperative Quality of Life Following Conventional Endodontic Intracanal Irrigation Compared with Laser-Activated Irrigation: A Randomized Clinical Study. Photobiomodul Photomed Laser Surg. 2019 Apr;37(4):248-253. doi: 10.1089/photob.2018.4558. PMID 31050955
- [Background] Topcuoglu HS, Topcuoglu G, Arslan H. The Effect of Different Irrigation Agitation Techniques on Postoperative Pain in Mandibular Molar Teeth with Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2018 Oct;44(10):1451-1456. doi: 10.1016/j.joen.2018.06.008. Epub 2018 Aug 23. PMID 30144989